CLINICAL TRIAL: NCT05543785
Title: Ketorolac for Intravenous Regional Analgesia in Lower Limb Orthopedic Surgeries Under Spinal Anesthesia: A Randomized Control Study
Brief Title: Ketorolac Intravenous Regional Analgesia in Lower Limb Surgeries
Acronym: K-IVRAg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R.22.09.1832
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain, Acute
Keywords: ketorolac; randomized controlled trial; intravenous regional anesthesia; lower limb; orthopedic surgeries
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Sodium Chloride; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: An anesthetist, not involved in the study, was responsible for randomization list construction, in blocks, opening the sealed envelopes and so, the preparation of the study drugs. The patient and the data collectors (anesthesia resident) does not know the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): will receive 50 ml normal saline in the intravenous regional cannula in the surgical limb with torniquet.
  And receive intravenous 30 mg ketorolac diluted in 10 ml saline in the peripheral general circulation.
  Interventions: Other: Control
- ketorolac (Active Comparator): will receive 15 mg ketorolac tromethamine diluted in normal saline in a total volume of 50 ml in the intravenous regional cannula in the surgical limb with torniquet.
  And receive intravenous 10 ml saline in the peripheral general circulation.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — After confirmation of circulatory isolation of the operated limb by the inflated tourniquet, 30 mg ketorolac tromethamine diluted in normal saline in a total volume of 50 ml will be injected
  Other Names: ketolac; Toradol; Biorolac
  Arms: ketorolac
Other: Control — After confirmation of circulatory isolation of the operated limb by the inflated tourniquet, 50 ml normal saline without drugs will be injected
  Other Names: Saline without drugs
  Arms: control

SUMMARY:
Tourniquet, a compressing device, otherwise its use in intravenous regional anesthesia, is commonly used in particular orthopedic surgeries. From the previous documented effectiveness and safety of intravenous (IV) administration of ketorolac in the circulatory-isolated limb as a part of intravenous regional anesthesia; we hypothesized that in orthopedic surgeries done with tourniquet, intravenous (IV) administration of ketorolac after tourniquet inflation, will act as intravenous regional analgesia. So, it will prolong the postoperative analgesic duration as a primary outcome.

DETAILED DESCRIPTION:
This is a randomized controlled trial that tests the effecacy of the intravenous regional ketorolac in lower limb orthopedic surgeries with spinal anesthesia. The investigators will compare the effect of 30 mg ketorolac without local anesthetic in the injected intravenously in an isolated lower limb (with torniquet) versus intravenous 30 mg ketorolac administered 10 minutes before toniquet pressuerization on the postoperative analgesia.

All patients will receive spinal anesthesia aiming for at least T12-L1 level. Postoperative standard analgesia will be paracetamol and diclofenac, given for both groups.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II
* Elective unilateral lower limb orthopedic surgery with tourniquet under spinal anesthesia

Exclusion Criteria:

* Pregnant females
* Body mass index ≥ 35 kg/m2
* Allergy to ketorolac
* Had renal, asthmatic, vascular (Raynaud's syndrome) disease, hematological anemias
* Had any history of gastrointestinal tract inflammation, bleeding, ulceration, or perforation besides
* Edema in the operated limb grade ≥ 3

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The postoperative analgesic duration | within 24 hours after the surgery
  the time measured from the onset of spinal anesthesia to the first request of analgesia by the patient

SECONDARY OUTCOMES:
Postoperative pain at rest | at 2, 4, 6, 12, 24 hours after 24 hours after surgery
  0-10 centimetres visual analog scale (VAS) for pain, where zero is equal to no pain and ten indicates the worst possible pain.
Postoperative pain at movement | at 2, 4, 6, 12, 24 hours after 24 hours after surgery
  0-10 centimetres visual analog scale (VAS) for pain, where zero is equal to no pain and ten indicates the worst possible pain. Movement will be standardized as 10 cm elevation of the surgical limb off the bed.
Total postoperative analgesic consumption | within the first 24 hours after surgery
  total amount of fentanyl as requested by the patient
time to sensory recovery from spinal anesthesia | through the intraoperative or postoperative care unit
  time to receovery of pin brick sensation at S1
time to motor recovery from spinal anesthesia | through the intraoperative or postoperative care unit
  time to modified Bromage score 0

OTHER OUTCOMES:
superficial vnous thrombophilibitis | intraoperative period
  redness or warmth noted at the proximal course of the injected vein before sterilization for surgery and at the end of surgery
postoperative bleeding tendency | over the first 24 hours after surgery
  the amount of the wound drain
wound healing | postoperative till the time to remove all wound sutures
  time to all wound sutures removed

CONTACTS AND LOCATIONS:
Overall Officials: Maha AboZeid, MD, Study Director — Mansoura University, Faculty of Medicine -
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Egypt